CLINICAL TRIAL: NCT02204514
Title: The Effects of Surgery for Painful External Snapping Hip
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Principal Investigator, Ole Simonsen, MD, DMSc, Northern Orthopaedic Division, Denmark
Other Study IDs: Surgery for ext. snapping hip
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Hip Pain
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery for external snapping hip
  Interventions: Procedure: Surgery for external snapping hip

INTERVENTIONS:
Procedure: Surgery for external snapping hip

SUMMARY:
The purpose of this study is to assess the pain-relieving effects of surgery for painful external snapping hip.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for painful external snapping hip
* 18 years or older

Exclusion Criteria:

* Inability to comply with the protocol (e.g. due to dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery for painful external snapping hip in The North Denmark Region between 2008-2013 with at least 1 year follow-up time.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | 1-6 years after surgery
  Do you still have the same pain as before surgery? Response categories: yes; no

CONTACTS AND LOCATIONS:
Overall Officials: Søren T Skou, PT, MSc, Principal Investigator — Orthopedic Surgery Research Unit + Department of Health Science and Technology, Aalborg University; Stine Jorstad, BSc, Study Chair — Department of Orthopedic Surgery; Ole Simonsen, MD, DMSc, Study Chair — Department of Orthopedic Surgery; Anders C Laursen, MD, Study Chair — Department of Orthopedic Surgery; Michael Ulrich, MD, PhD, DMSc, Principal Investigator — Department of Orthopedic Surgery
Locations (1):
- Department of Orthopedic Surgery, Aalborg, Denmark